CLINICAL TRIAL: NCT06071273
Title: Development of an Online Platform for Self-service of People Living With Chronic Cardiovascular Diseases
Brief Title: Online Platform for Self-service of Patients With Chronic Cardiovascular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evangelia Kouidi, Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ΚΜΡ6-0076626
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home-based exercise (Experimental): 6 months home-based exercise program with continuous monitoring of the cardiovascular response of the participants during exercise via the online platform.
  Interventions: Other: Group A: online real-time home based exercise using the online platform
- Community-based exercise (Experimental): 6-month community based (i.e., local community gym) exercise intervention
  Interventions: Other: Group B: supervised community based exercise intervention
- Control group (No Intervention): Control group, no exercise intervention.

INTERVENTIONS:
Other: Group A: online real-time home based exercise using the online platform — Patients that will be randomly assigned to this group will be exercising at home by providing data of their vital signs during exercise and at rest. To succeed this, they will be provided with the appropriate equipment (e.g., a smart watch able to assess the electrical signs of the heart (i.e., ECG) and heart rate, an automated blood pressure monitor, and an electrical body scale) which will be directly linked to the online platform.
  The online real-time supervised home-based exercise program is identical to Group B, the only difference is that it is performed at home. Each session has a duration of 60 minutes consisting of 40 mins of aerobic exercise and 20mins of resistance training. The overall intensity is kept to moderate based on ratings of perceived exertion (i.e., 13-14 in Borg's scale 6-20). The program will last for 6 months with exercise sessions taking place thrice per week.
  Arms: Home-based exercise
Other: Group B: supervised community based exercise intervention — Identical exercise program to Group A, the only difference is that Group performs the supervised exercise in community based health clubs/gyms.
  Arms: Community-based exercise

SUMMARY:
The purpose of this study is to define the requirements and characteristics of the software that will be developed for the project "Creation of a platform for self-service of people living with chronic cardiovascular diseases in an understandable, clear, complete, consistent and verifiable manner.

The project concerns the design and implementation of a long-term program of therapeutic exercise and evaluation, by exercise and health professionals, of the anatomical and functional adaptations of exercise in patients and athletes with cardiovascular diseases. Essentially, it is a program of recording and monitoring cardiovascular rehabilitation in the form of systematic exercise of the patient both at home and in sports venues, which will contribute to the prevention of cardiovascular events in conditions of fatigue and at rest as well as to the gradual rehabilitation of the patient who performs a physical activity.

Depending on the individual's functional capacity and health issues, combined with monitoring the patient's vital signs (such as blood pressure, heart rate, oxygen saturation, body temperature) the exercise professional will create an individualized, targeted exercise program with ultimate aiming at its rehabilitation with the help of physical activity and the improvement of its functional performance and by extension the quality of life of the individual. At the same time, the project will seek to motivate patients to remain committed to the physical activity program, with the aim of faster reintegration into their daily life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiovascular disease and recent myocardial infarction (>4weeks)
* Patients shall be in a clinical stable condition.

Exclusion Criteria:

* Uncontrolled T1 or T2 diabetes mellitus.
* Comorbidities precluding exercise training (e.g., orthopaedic/neurological conditions).
* Uncontrolled arrhythmias

Ages: 40 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Physical activity levels | 6 months
  Physical activity levels will be assessed by mean daily step count for all groups including the control group.

SECONDARY OUTCOMES:
Cardiorespiratory fitness (CRF) | 6 months
  CRF will be assessed by performing a peak oxygen uptake test at baseline and post-exercise intervention for all groups including the control group.
Percentage of body fat mass | 6 months
  Body composition analysis will be performed via bioelectrical impedance to assess the levels of fat (%) pre and the intervention for all groups, including the control group.
Body muscle mass | 6 months
  Body composition analysis will be performed via bioelectrical impedance to assess the levels of muscle mass (kg) pre and the intervention for all groups, including the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Thermi, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitropoulos A, Anifanti Mu, Koukouvou G, Ntovoli Alpha, Alexandris K, Kouidi E. Exploring the feasibility, acceptability, and safety of a real-time cardiac telerehabilitation and tele coaching programme using wearable devices in people with a recent myocardial infarction. BMC Sports Sci Med Rehabil. 2024 Sep 30;16(1):207. doi: 10.1186/s13102-024-00992-5. PMID 39350291